CLINICAL TRIAL: NCT06644209
Title: Predictive Efficacy of Ratio of Median Frequency to Spectral Edge Frequency Used in the Depth of Anaesthesia Monitoring on Post-operative Cognitive Functions
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Basak Ceyda MECO, Prof. Dr., Ankara University
Other Study IDs: AU-BY-001
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Postoperative Delirium; Cognitive Impairment
Keywords: Bispectral Index; Median Frequency; Spectral Edge Frequency; Post Operative Cognitive Dysfunction; Cognition
MeSH Terms: conditions — Emergence Delirium; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The primary objective of this observational study is to evaluate the effectiveness of preoperative anaesthesia depth monitoring parameters in predicting postoperative cognitive functions in non-cardiac adult patients.

Participants will preoperatively perform cognitive tests such as the Nursing Delirium Screening Scale(Nu-DESC) and 4 'A's Test(4AT) to assess baseline cognitive performance. The same tests will be repeated twice daily until the postoperative 3rd day or discharge.

DETAILED DESCRIPTION:
The primary objective of this observational study is to evaluate the effectiveness of preoperative anaesthesia depth monitoring parameters such as Bispectral Index(BIS), Spectral edge frequency(SEF) and Median frequency(MF) in predicting postoperative cognitive functions in non-cardiac adult patients.

Participants will preoperatively perform cognitive tests such as the Nursing Delirium Screening Scale(Nu-DESC) and 4 'A's Test(4AT) to assess baseline cognitive performance. Intraoperative haemodynamic and BIS parameters will be collected via manual data entry into printed forms. Also, a two-channel electroencephalogram(EEG) and BIS parameters(BIS Number, SEF, MF) will be collected digitally.

The cognitive tests will be repeated twice daily until the postoperative 3rd day or discharge.

Parameters such as mean intraoperative MF value and the ratio of MF over SEF will be compared against postoperative cognitive test scores.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (aged over 18 years), Patients undergoing elective surgeries, Patients consenting to participate in the study.

Exclusion Criteria:

Pediatric patients (aged under 18 years), Patients undergoing emergency surgeries, Patients requiring or anticipated to require postoperative intensive care for more than one day, Patients undergoing cardiac surgeries, Patients undergoing intracranial surgeries, Patients are undergoing endoscopic sinus or brain surgeries, Patients with pacemakers or implantable cardioverter-defibrillators (ICDs), Patients diagnosed with dementia (including Alzheimer's disease, Lewy body dementia, etc.), Patients with chronic opioid or benzodiazepine use, Patients with contraindications to Propofol, Remifentanil, or Fentanyl, Pregnant or breastfeeding women, Patients are not willing to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The research focuses on adults (≥18 years old) of any gender residing in Türkiye, scheduled for elective, non-cardiac surgeries.
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2024-01-25 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Nu-DESC Score | 3 Days
  Increase in Nu-DESC score compared to baseline test, or a postoperative Nu-DESC score greater than or equal to 2
4AT Score | 3 Days
  Increase in 4AT score compared to baseline test, or a postoperative 4AT score greater than or equal to 4

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koch S, Windmann V, Chakravarty S, Kruppa J, Yurek F, Brown EN, Winterer G, Spies C; BioCog Study Group. Perioperative Electroencephalogram Spectral Dynamics Related to Postoperative Delirium in Older Patients. Anesth Analg. 2021 Dec 1;133(6):1598-1607. doi: 10.1213/ANE.0000000000005668. PMID 34591807